CLINICAL TRIAL: NCT01130948
Title: Sleep, Breathing and Psychomotor Performance at Altitude: A Physiologic Study in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 2010-0054/1
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Healthy Men
Keywords: hypoxia; altitude; sleep; sleep apnea; periodic breathing; vigilance; psychomotor; endothelial function
MeSH Terms: conditions — Hypoxia; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: altitude exposure — exposure to 490m, 1700m and 2590m

SUMMARY:
This study investigates the effect of altitude exposure on sleep, breathing and psychomotor performance in healthy subjects.

DETAILED DESCRIPTION:
Sleep is essential for well being and performance. Sleep disturbances by recurrent apnea and hypoxia in patients with obstructive sleep apnea syndrome impair quality of life, cognitive and cardiovascular functions. Similar consequences occur in healthy subjects exposed to hypoxia at altitude due to periodic breathing with recurrent central apnea. This project will investigate effects of altitude on sleep, breathing, psychomotor performance and on the cardiovascular system in healthy subjects and patients with sleep apnea. The results will help to better understand mechanisms of sleep disturbances and psychomotor impairment induced by hypoxia and to prevent adverse effects of altitude exposure.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* residence at <800m

Exclusion Criteria:

* any active disease requiring treatment
* requirement for regular use of medication
* smoking, regular intake of alcohol or drugs
* body mass index <18 or >30 kg/m2
* previous intolerance of moderate altitude (<3000m)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
apnea/hypopnea index | day 1-4 at altitude
Reaction time | day 1-4 at altitude
  psychomotor vigilance test reaction time

SECONDARY OUTCOMES:
Psychomotor vigilance | day 1-4 at altitude
  performance in the Motor Task Manager test
sleep quality | day 1-4 at altitude
  percent of slow wave sleep, araousal index
arterial applanation tonometry | day 1-4 at altitude
  endothelial function and arterial stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, Prof. MD, Principal Investigator — University Hospital Zurich, Pulmonary Division
Locations (1):
- University Hospital of Zurich, Pulmonary Division, Zurich, Switzerland

REFERENCES:
- [Background] Latshang TD, Lo Cascio CM, Stowhas AC, Grimm M, Stadelmann K, Tesler N, Achermann P, Huber R, Kohler M, Bloch KE. Are nocturnal breathing, sleep, and cognitive performance impaired at moderate altitude (1,630-2,590 m)? Sleep. 2013 Dec 1;36(12):1969-76. doi: 10.5665/sleep.3242. PMID 24293773
- [Background] Stadelmann K, Latshang TD, Tarokh L, Lo Cascio CM, Tesler N, Stoewhas AC, Kohler M, Bloch KE, Huber R, Achermann P. Sleep respiratory disturbances and arousals at moderate altitude have overlapping electroencephalogram spectral signatures. J Sleep Res. 2014 Aug;23(4):463-8. doi: 10.1111/jsr.12131. Epub 2014 Feb 19. PMID 24552365
- [Background] Ayers L, Stoewhas AC, Ferry B, Latshang TD, Lo Cascio CM, Sadler R, Stadelmann K, Tesler N, Huber R, Achermann P, Bloch KE, Kohler M. Circulating levels of cell-derived microparticles are reduced by mild hypobaric hypoxia: data from a randomised controlled trial. Eur J Appl Physiol. 2014 May;114(5):1067-73. doi: 10.1007/s00421-014-2837-6. Epub 2014 Feb 11. PMID 24514947
- [Background] Stadelmann K, Latshang TD, Lo Cascio CM, Tesler N, Stoewhas AC, Kohler M, Bloch KE, Huber R, Achermann P. Quantitative changes in the sleep EEG at moderate altitude (1630 m and 2590 m). PLoS One. 2013 Oct 22;8(10):e76945. doi: 10.1371/journal.pone.0076945. eCollection 2013. PMID 24167552
- [Background] Stowhas AC, Latshang TD, Lo Cascio CM, Lautwein S, Stadelmann K, Tesler N, Ayers L, Berneis K, Gerber PA, Huber R, Achermann P, Bloch KE, Kohler M. Effects of acute exposure to moderate altitude on vascular function, metabolism and systemic inflammation. PLoS One. 2013 Aug 1;8(8):e70081. doi: 10.1371/journal.pone.0070081. Print 2013. PMID 23936377
- [Derived] Stadelmann K, Latshang TD, Lo Cascio CM, Clark RA, Huber R, Kohler M, Achermann P, Bloch KE. Impaired postural control in healthy men at moderate altitude (1630 m and 2590 m): data from a randomized trial. PLoS One. 2015 Feb 27;10(2):e0116695. doi: 10.1371/journal.pone.0116695. eCollection 2015. PMID 25723529